CLINICAL TRIAL: NCT01649505
Title: Intraoperative Use of Fibrin Glue Sealant Combined With Sharp Dissection Technique as a Preventative Measure for Seromas
Brief Title: Fibrin Sealant in Preventing Fluid Build Up During Surgery in Patients Undergoing Breast Reconstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low patient enrollment and no clinical findings.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Juliana Hansen, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00006606; NCI-2012-00809 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Perioperative/Postoperative Complications
MeSH Terms: conditions — Breast Neoplasms; Postoperative Complications | interventions — Fibrin Tissue Adhesive; Mammaplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (fibrin sealant) (Experimental): Patients undergo sharp dissection technique with fibrin sealant closure.
  Interventions: Drug: fibrin sealant (Beriplast P, TISSEEL VH); Procedure: breast reconstruction
- Arm II (standard electrocoagulation) (Active Comparator): Patients undergo standard electrocoagulation dissection technique.
  Interventions: Procedure: breast reconstruction

INTERVENTIONS:
Drug: fibrin sealant (Beriplast P, TISSEEL VH) — Applied topically
  Other Names: Beriplast P; TISSEEL VH
  Arms: Arm I (fibrin sealant)
Procedure: breast reconstruction — Undergo sharp dissection technique
  Other Names: Mammaplasty
  Arms: Arm I (fibrin sealant)
Procedure: breast reconstruction — Undergo electrocoagulation dissection technique
  Other Names: Mammaplasty
  Arms: Arm II (standard electrocoagulation)

SUMMARY:
The purpose of this study is to investigate the efficacy of an alternative surgical technique and the use of fibrin sealant in preventing post-operative seroma formation. A seroma is a build-up of clear bodily fluids in a place on the body where tissue has been removed by surgery. Seromas can happen after breast surgeries. Seromas can appear about 7 to 10 days after surgery, after the drainage tubes have been removed. The breast area involved in the surgery may have a spot that's swollen and feels like there is liquid under the skin

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate differing surgical techniques (sharp dissection v. electrosurgical, use of fibrin glue) in latissimus dorsi donor flap harvest and their effect, if any on the prevention of post-operative seromas.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo sharp dissection technique with fibrin sealant closure.

ARM II: Patients undergo standard electrocoagulation dissection technique.

After completion of study treatment, patients are followed up for 90-180 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be undergoing latissimus dorsi donor flap harvest reconstruction and evaluated by the Department of Plastic and Reconstructive Surgery at Oregon Health and Science University (OHSU)
* These patients will be undergoing reconstructive surgery for a mastectomy/wide local excision of breast cancer defect or other soft tissue defect resulting from trauma, infection, undesirable surgical outcome, oncologic resection, etc.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who will not qualify for latissimus dorsi donor flap reconstruction based on anatomical limitations specific the subjects respectively; to be evaluated by the plastic surgeon
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fibrin glue sealant
* Patients with evidence of hematological disorders resulting in deficient coagulation whereby sharp dissection would result in undesirable bleeding otherwise performed more safely with electrosurgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Hansen, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Fibrin Sealant): Patients undergo sharp dissection technique with fibrin sealant closure.
  breast reconstruction : Undergo sharp dissection technique
  fibrin sealant (Beriplast P, TISSEEL VH) : Applied topically
- Arm II (Standard Electrocoagulation): Patients undergo standard electrocoagulation dissection technique.
  breast reconstruction : Undergo electrocoagulation dissection technique
Period: Overall Study
Arm/Group | Arm I (Fibrin Sealant) | Arm II (Standard Electrocoagulation)
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Fibrin Sealant) | Arm II (Standard Electrocoagulation) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 | 44 | 44 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in Each Arm Who Develop Post-operative Seromas
Description: Computed with 95% confidence interval using exact method. The difference of seroma rate in the two groups will be computed with 95% confidence interval using exact method. Two-sided Fisher's exact test will be used to evaluate whether the seroma rate are significantly different for the two treatment groups.
Time Frame: Up to day 180 post-operation
Population: Data was not collected due to early termination and very low accrual
Arm/Group | Arm I (Fibrin Sealant) | Arm II (Standard Electrocoagulation)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Patients Who Experienced Wound Infections, Wound Separation, or Any Other Surgical Complications
Description: Computed with 95% confidence interval using exact method. Two-sided Fisher's exact test will be used to evaluate whether the wound complication rate are significantly different for the two treatment groups, and the odds ratio with 95% confidence interval will be computed.
Time Frame: Up to day 180 post-operation
Population: Data was not collected due to early termination and very low accrual
Arm/Group | Arm I (Fibrin Sealant) | Arm II (Standard Electrocoagulation)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quantity of Post-operative Drainage
Description: Defined as total volume of drainage recorded (in ml) by nurses while the patient is in the hospital and by patient himself/herself when discharged home, until the removal of the drain by a doctor once it reaches less than 50 ml per day. Wilcoxon rank sum test will be used to compare the drainage volume of the two groups.
Time Frame: Up to day 10 post-operation
Population: Data was not collected due to early termination and very low accrual
Arm/Group | Arm I (Fibrin Sealant) | Arm II (Standard Electrocoagulation)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Serious and Nonserious Adverse Events and Complications
Time Frame: Up to day 180 post-operation
Population: Data was not collected due to early termination and very low accrual
Arm/Group | Arm I (Fibrin Sealant) | Arm II (Standard Electrocoagulation)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Fibrin Sealant) | Arm II (Standard Electrocoagulation)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Data was not collected due to early termination and very low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes